CLINICAL TRIAL: NCT05881694
Title: Accuracy of Combined Upper Lip Bite Test and Ultrasound Measurement of Skin-to-epiglottis Distance in Predicting Difficult Laryngoscopy: a Prospective Observational Study
Brief Title: Accuracy of Upper Lip Bite Test and Measurement of Skin-to-epiglottis Distance in Predicting Difficult Laryngoscopy: a Prospective Observational Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sherin Refaat, Assisstant professor of anesthiology ,faculty of medcine ,Cairo univeristy, Cairo University
Other Study IDs: MS-122-2022
Record Dates: First submitted 2023-05-21; First posted 2023-05-31 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-06

CONDITIONS: Difficult Laryngoscopy; Upper Lip Bite Test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Airway management is one of the most important skills in everyday practice of anesthesia. Improper airway management might lead to high risk of mortality. clinical parameters alone cannot predict all potentially difficult airways. Ultrasonography (US) might play a role as a potential screening tool for difficult airway and given the limited empirical study in this field; this research will focus on using ultrasound to predict difficult airway and difficult mask ventilation for patients undergoing elective operation under general anesthesia. Methodology This study is Prospective observational . The study will be conducted in Cairo University Hospital Participants are adult patients (above >40 years), (BMI < 35) with American Society of Anesthesiologists physical status (ASA-PS) I-III, scheduled for elective surgery under general anesthesia with tracheal intubation . Exclusion criteria included patients with history of difficult intubation or apparent airway abnormalities (facial scars, neck scars, unstable cervical spine and history of cervical spine fixation) that would require alternative technique other than endotracheal intubation with direct laryngoscopy. Also, edentulous patients, patients undergoing emergency procedure and pregnant women are excluded from the study. Hypothesis The investigators hypothesize that combined class 3 ULBT and DSE >2 cm can accurately predict difficult laryngoscopy in adult patients undergoing elective procedure under general anesthesia with endotracheal intubation.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be adult patients (above >40 years) ( BMI < 35) with ASA-PS I-III, scheduled for elective surgery under general anesthesia with tracheal intubation.

Exclusion Criteria:

* Patients with history of difficult intubation or apparent airway abnormalities (facial scars, neck scars, unstable cervical spine and history of cervical spine fixation) that would require alternative technique other than endotracheal intubation.

Edentulous patients patients undergoing emergency procedure pregnant women were excluded from the study.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: adult patients (above >40 years) ,( BMI < 35) with ASA-PS I-III, scheduled for elective surgery under general anesthesia with tracheal intubation
Sampling Method: Non-Probability Sample
Enrollment: 210 (Estimated)
Dates: Start 2023-05-30 (Estimated); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-10-05 (Estimated)

PRIMARY OUTCOMES:
The accuracy of combined class 3 ULBT and DSE >2 cm in predicting difficult laryngoscopy | before start of anesthesia till intubation of the patient
  The ULBT was performed by asking the patient to bite their upper lip with the lower incisors as high as they could While the patient was in supine position with the head in neutral position, the transducer was placed in the transverse plane at the level of the thyrohyoid membrane. The epiglottis was visible through the thyrohyoid membrane as a hypoechoic curvilinear structure with its posterior border demarcated by a bright hyperechoic linear air-mucosal interface. For each patient, the distance from the skin to the epiglottis was measured three times at the central axis of the epiglottis and the average of the measurement was calculated.